CLINICAL TRIAL: NCT02310178
Title: Obesity Cohort : Medical Follow-up of Severe or Morbid Obese Patients Undergoing Bariatric Surgery
Acronym: BAREVAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UF 8855
Record Dates: First submitted 2014-10-28; First posted 2014-12-08 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate
Keywords: weight loss; sleeve gastrectomy; gastric bypass; gastric banding; bariatric procedures; cohort; morbid obesity; medical and economical impact; severe obesity
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group/Cohort (Other): all of the current bariatric surgeries are allowed in this prospective cohort study
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — all of the current bariatric surgeries are allowed in this prospective cohort study

SUMMARY:
The aim of this cohort is to evaluate the follow-up of morbidly obese patients treated by several types of bariatric procedures. In addition, this study could lead to the development of clinical trials on assessment of the bariatric surgery impact.

DETAILED DESCRIPTION:
The main objective is to prospectively evaluate long-term efficiency of bariatric surgery in terms of weight loss. Moreover, this cohort wants to assess the long-term effectiveness of bariatric surgery on comorbidities and quality of life, the medical and economic impact of bariatric surgery (before-after comparison using data from health insurance), estimates the incidence of mortality and morbidity of bariatric surgery and to finish describe the evolution of patients in case of new-surgery. From a methodological point of view, the Obesity cohort is a prospective cohort study, single-center, open, with aftercare performed during life of patients. The number of inclusions is to 1500 patients. After surgery , patients will be followed at least 4 visits the first year and at least 2 visits a year then. The recommendations of the french health ministry (HAS), the frequency of visits may be increased according to the patient's progress. Follow-up visits of patients after bariatric surgery will be performed by physicians or surgeons of the multidisciplinary team responsible for the care of the patient (digestive and reconstructive surgery, anesthesiology, endocrinology, medical imaging, gastroenterology, immunology and physiology) . It will be insured for life, obesity is a chronic disease and because of the risk of late complications.

ELIGIBILITY:
Inclusion Criteria:

* Only be considered in patients operated and followed at CHU Montpellier with bariatric surgery
* Patients treated by bariatric surgery on CHU Montpellier
* Agreed to participate to the study by signing an informed consent
* Eligible to health insurance

Exclusion Criteria:

* Unable to follow the patient in the long term (foreign patients, surgical use ...)
* Inability to follow in the long run

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2012-05-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the long-term efficiency of bariatric surgery on weight loss | Change from intervention to 5 years
  Assessment of weight loss

SECONDARY OUTCOMES:
Assessment of the long-term efficiency of bariatric surgery on diabetes | Change from intervention to 5 years
  Assessment of blood glucose, HbA1c and diabetes medications
Assessment of the long-term efficiency of bariatric surgery on High Blood Pressure | Change from intervention to 5 years
  Assessment of Systolic Blood Pressure and blood pressure medications
Assessment of the long-term efficiency of bariatric surgery on dyslipidemia | Change from intervention to 5 years
  Assessment of cholesterolemia and triglyceridemia and dyslipidemia medications
Assessment of the long-term efficiency of bariatric surgery on rheumatism | Change from intervention to 5 years
  Assessment of rheumatism medications
Assessment of the long-term efficiency of bariatric surgery on respiratory pathologies | Change from intervention to 5 years
  Assessment of respiratory pathologies medications
Assessment of the long-term efficiency of bariatric surgery on sleep apnea syndrome | Change from intervention to 3 months
  polysomnography tests
Assessment of the long-term efficiency of bariatric surgery on quality of life | Change from intervention to 5 years
  Assessment of quality of life questionnaires (SF36 and BAROS)
Assessment of medico-economic impact of bariatric surgery | Change from intervention to 5 years
  Comparison of health insurance data
Assessment of mortality of bariatric surgery | Change from intervention to 5 years
  Assessment of the date of death

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU - Hôpital Saint Eloi, Montpellier, France

REFERENCES:
- [Derived] Saux P, Bauvin P, Raverdy V, Teigny J, Verkindt H, Soumphonphakdy T, Debert M, Jacobs A, Jacobs D, Monpellier V, Lee PC, Lim CH, Andersson-Assarsson JC, Carlsson L, Svensson PA, Galtier F, Dezfoulian G, Moldovanu M, Andrieux S, Couster J, Lepage M, Lembo E, Verrastro O, Robert M, Salminen P, Mingrone G, Peterli R, Cohen RV, Zerrweck C, Nocca D, Le Roux CW, Caiazzo R, Preux P, Pattou F. Development and validation of an interpretable machine learning-based calculator for predicting 5-year weight trajectories after bariatric surgery: a multinational retrospective cohort SOPHIA study. Lancet Digit Health. 2023 Oct;5(10):e692-e702. doi: 10.1016/S2589-7500(23)00135-8. Epub 2023 Aug 29. PMID 37652841
- [Derived] Nocca D, Galtier F, Taleb S, Picot MC, Jaussent A, Silvestri M, Lefebvre P, de Jong A, Gautier T, Loureiro M, Nedelcu M. Peri-operative Morbidity of Nissen Sleeve Gastrectomy: Prospective Evaluation of a Cohort of 365 Patients, Beyond the Learning Curve. Obes Surg. 2022 Jul;32(7):1-7. doi: 10.1007/s11695-022-06066-0. Epub 2022 May 7. PMID 35524904